CLINICAL TRIAL: NCT04655872
Title: A Phase I Study of the Mass Balance of a Single Oral Administration of [14C]TPN171H in Healthy Male Subjects
Brief Title: Mass Balance of Oral [14C]TPN171H in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vigonvita Life Sciences (Industry)
Collaborators: Shanghai Institute of Materia Medica, Chinese Academy of Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TPN171H-07
Record Dates: First submitted 2020-11-23; First posted 2020-12-07 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2020-11

CONDITIONS: Healthy Male Subjects
Keywords: Mass balance; TPN171H; Simmerafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]TPN171H (Experimental)
  Interventions: Drug: [14C]TPN171H

INTERVENTIONS:
Drug: [14C]TPN171H — A single 10 mg oral dose of [14C]TPN171H containing approximately 100 microcurie of [14C]-TPN171H.

SUMMARY:
This study is objective to evaluate the in vivo absorption, excretion and biotransformation pathways of [14C]-TPN171H in Chinese male healthy volunteers, and to reveal the overall pharmacokinetic characteristics of TPN171H in human body, so as to provide basis for rational use of the drug.

DETAILED DESCRIPTION:
This will be an open-label, single-center study to evaluate the mass-balance and pharmacokinetics of TPN171H in approximately 6 healthy male subjects receiving a single oral 10 mg dose of TPN171H containing approximately 100 microcuries of [14C]-TPN171H. Subjects will be checked in to the research unit from approximately 24 hours prior to dosing and remain in house until greater than 80% of the administered radioactivity is collected from bodily excreta or until less than 1% of the administered radioactivity is recovered from excreta in two consecutive time intervals, and blood sample radioactivity concentration at two consecutive time points less than 3 times the plasma background value. This study will investigate the main biotransformation and elimination pathways of TPN171H in the human body and will seek to identify compound's major metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 19 and 55 years,with normal bowel movements (1~2 times a day);
* Body Mass Index of 19 to 26 kg/m2; Body weight no less than 50 kg;
* Physical examination, vital signs examination, laboratory examination (blood routine, urine routine, blood biochemistry, thyroid function, stool routine and occult blood, etc.), 12 lead ECG, B-ultrasound, chest X-ray and fundus examination results were normal or abnormal without clinical significance;
* The male subjects with fertility had no child rearing plan or sperm donation plan with their sexual partners during the trial and within one year after taking the drug, and could take reliable contraceptive measures;
* Fully understand the purpose and requirements of this trial, voluntarily participate in the clinical trial and sign the written informed consent, and can complete the whole trial process according to the test requirements.

Exclusion Criteria:

* People with allergies or allergic diseases, or known allergies to test preparations, any of their ingredients, and related preparations;
* There are clear diseases of the central nervous system, cardiovascular system, digestive system (including those with severe fatty liver in B-ultrasound examination), respiratory system, urinary system, blood system, metabolic disorders, etc. and require medical intervention or other unsuitable clinical trials Those with tested diseases (such as history of mental illness, etc.); those with a history of orthostatic hypotension;
* Blurred vision or a history of the following ocular diseases: nonvascular anterior ischemic optic neuropathy (NAION), abnormal color vision, hereditary retinal degeneration (such as retinitis pigmentosa), macular degeneration;
* Any drug that inhibits or induces liver drug-metabolizing enzymes (inducers-barbiturates, carbamazepine, phenytoin, rifampicin, dexamethasone, rifabutin, rifapentine) has been used within 30 days before administration ; Inhibitors-SSRI antidepressants, cimetidine, diltiazem, macrolides, verapamil, imidazole antifungals, sedatives and hypnotics, fluoroquinolones, antihistamines, etc.);
* Those who have taken any prescription drugs, over-the-counter drugs, Chinese herbal medicines or health care products within 2 weeks before administration; or those who have participated in other drug clinical trials and received trial drugs within 3 months before administration;
* Those who have a history of drug dependence (including a history of drug use) within 2 years before administration; or urine drug abuse screening (morphine, tetrahydrocannabinol acid, methamphetamine, dimethylene oxyamphetamine) , Ketamine and cocaine) positive;
* Those who smoke more than 10 cigarettes per day and do not agree to avoid using any tobacco products during the trial period;
* Positive results of alcohol breath test, or current/previous alcoholics (drinking more than 21 standard units per week. 1 standard unit contains 14 g of alcohol, such as 360 mL of beer or 45 mL of 40% spirits or 150 mL wine);
* People who have consumed excessive amounts of grapefruit juice, tea, coffee and/or caffeinated beverages for a long time (more than 8 cups a day, 1 cup equal to 250 mL);
* Those who are positive for hepatitis B surface antigen (HBsAg), HCV antibody, syphilis antibody and HIV antibody;
* Blood loss or blood donation of 400 mL or more within 3 months before administration;
* Those who have been vaccinated within 6 months before administration;
* A history of fainting needles or fainting blood;
* Hemorrhoids or perianal diseases with regular/current stools; habitual constipation or diarrhea, irritable bowel syndrome, inflammatory bowel disease;
* Workers who need to be exposed to radioactive conditions for a long time; or have significant radioactive exposure more than 2 chest/abdominal CT, or more than 3 other types of X-ray examinations) within 1 year before administration or participated in radiopharmaceutical labeling Experimenter
* The investigator believes that there are other factors that are not suitable for participating in this trial.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2020-11-26 (Actual); Primary Completion 2021-01-27 (Actual); Study Completion 2021-01-27 (Actual)

PRIMARY OUTCOMES:
Cmax - maximum observed plasma concentration | From time zero up to 336 hours post-dose following oral administration of [14C]TPN171H
Tmax - time at which Cmax occurs | From time zero up to 336 hours post-dose following oral administration of [14C]TPN171H
AUC0~t - area under the plasma concentration time curve from time zero to the last measurable concentration | From time zero up to 336 hours post-dose following oral administration of [14C]TPN171H
AUC0-∞ - area under the plasma concentration-time curve from time zero to infinity | From time zero up to 336 hours post-dose following oral administration of [14C]TPN171H
Total radioactivity in urine and faeces | From time zero up to 336 hours post-dose following oral administration of [14C]TPN171H

CONTACTS AND LOCATIONS:
Overall Officials: Gangyi Liu, Principal Investigator — Shanghai Xuhui Central Hospital
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No